CLINICAL TRIAL: NCT04840732
Title: Virtual Reality Application in Chemotherapy Administration in Nurse Staff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: VR for nurse
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-04

CONDITIONS: Chemotherapy Training
Keywords: 3D virtual reality; administration

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and Outcomes Assessor blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention (Experimental): The experimental group uses the VR program to training chemotherapy skill. Use VR software to make a training education program.
  Interventions: Behavioral: VR training program
- No Intervention: usual care (Placebo Comparator): Chemotherapy training as usual care (for training chemotherapy skill).
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: VR training program — Use VR software to make a training education program.
  Arms: Experimental: Intervention
Behavioral: usual care — Chemotherapy training as usual care (for training chemotherapy skill).
  Arms: No Intervention: usual care

SUMMARY:
The present study wants to design a training program for chemotherapy with using VR among nurse staff. Then the investigators design a protocol to compare the training effects in the VR program and ISO document.

DETAILED DESCRIPTION:
As technology advances, mobile devices have gradually turned into wearable devices. Furthermore, virtual reality (VR), augmented reality (AR), and mixed reality (MR) are being increasingly applied in medical fields such as medical education and training, surgical simulation, neurological rehabilitation, psychotherapy, and telemedicine. Research results demonstrate the ability of VR, AR, and MR to ameliorate the inconveniences that are often associated with traditional medical care, reduce incidents of medical malpractice caused by unskilled operations, and reduce the cost of medical education and training. What is more, the application of these technologies has enhanced the effectiveness of medical education and training, raised the level of diagnosis and treatment, improved the doctor-patient relationship, and boosted the efficiency of medical execution. The present study wants to design a training program for chemotherapy with using VR. Then the investigators design a protocol to compare the training effects in VR program and ISO document.

ELIGIBILITY:
Inclusion Criteria:

* The staffs who require to implement chemotherapy skill in the hospital. Age over 20 years.

Exclusion Criteria:

* Refuse to join the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Objective Structured Clinical Examination score (OSCE score) | One month
  One month after intervention, we assess the OSCE score from participates, range from 0 to 100, higher score means better grade.

SECONDARY OUTCOMES:
Self-assessment skill score | One month
  The confidence of Self-assessment skill score after intervention. Range from 0 to 100, higher score means better grade.

OTHER OUTCOMES:
Knowledge and attitude (pre test) | baseline data
  Chemotherapy knowledge and attitude, range 5-50, higer score means higher attitude to do chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei County, Taiwan

REFERENCES:
- [Derived] Wang CY, Lu CY, Yang SY, Tsai SC, Huang TW. 3D Virtual Reality Smartphone Training for Chemotherapy Drug Administration by Non-oncology Nurses: A Randomized Controlled Trial. Front Med (Lausanne). 2022 Jun 20;9:889125. doi: 10.3389/fmed.2022.889125. eCollection 2022. PMID 35795629